CLINICAL TRIAL: NCT02746822
Title: Thrombus Aspiration in Acute ST-elevation Myocardial Infarction
Acronym: TASTI
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Svein Solheim, MD, PhD, Oslo University Hospital
Other Study IDs: 2015/169
Record Dates: First submitted 2016-04-08; First posted 2016-04-21 (Estimated); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Acute ST-elevation Myocardial Infarction
Keywords: acute myocardial infarction,; thrombus aspiration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — thrombus material and blood
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other:

SUMMARY:
Thirty patients with acute ST-elevation myocardial infarction treated with primary PCI and aspiration of thrombus material from the infarct related coronary artery will be included. Both cellular and non cellular content of the thrombus will be examined with morphological and immunohistochemical methods and related to time from onset of symptoms to PCI, as well as to the degree of myocardial necrosis. Furthermore, mRNA expression of selected signal molecules will be performed. In addition, peripheral venous blood samples will be drawn and analyzed for signalling molecules and corresponding mRNA expression in circulating leukocytes.

DETAILED DESCRIPTION:
Observational, cross-sectional study on 30 patients with STEMI treated with thrombectomy and PCI with stent implantation. Composition and characteristics of the coronary thrombi with respect to cell types, genetic expression and presence of specific markers of inflammation, platelet activity, endothelial activation, coagulation and fibrinolysis will be investigated in relation to the levels of these markers in the general circulation, and specifically related to the time axis from symptom to PCI, as well as to the degree of myocardial necrosis.

Intracoronary thrombus will be retrieved by standard aspiration catheter, washed with saline and stored on formalin as advised by the Department of pathology, OUS Ullevål. A specific protocol for morphological and immunohistochemical methods is prepared and has been shown suitable in a pilot study on 5 patients. Assessment of coronary TIMI flow and peripheral blush grade after thrombus aspiration and PCI will be done. At the same time, peripheral venous blood will be drawn, processed and stored at -80˚C for later analyses. Demographic variables will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Both gender
* age 18-75 years
* typical symptoms of acute myocardial infarction
* ST-elevation or presumed new left bundle branch block in the ECG
* treated with aspiration of thrombus and primary PCI in the infarct related coronary artery

Exclusion Criteria:

* Signs of infection
* pulmonary embolism
* chronic obstructive pulmonary disease
* arrhythmias, abnormal renal and/or liver function
* autoimmune disease
* malignant disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute St-elevation myocardial infarction
Sampling Method: Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2015-04; Primary Completion 2019-01-09 (Actual); Study Completion 2019-01-09 (Actual)

PRIMARY OUTCOMES:
Cell composition of the intracoronary thrombus related to symptom length | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Ingebjørg Seljeflot, Professor, Study Chair — Kirkeveien 166, 0407 Oslo, Norway
Locations (1):
- Department of Cardiology, Oslo University Hospital, Ullevål, Oslo, Norway

REFERENCES:
- [Derived] Nordeng J, Solheim S, Akra S, Schandiz H, Hoffmann P, Roald B, Bendz B, Arnesen H, Helseth R, Seljeflot I. Gene expression of fibrinolytic markers in coronary thrombi. Thromb J. 2022 Apr 29;20(1):23. doi: 10.1186/s12959-022-00383-1. PMID 35488283
- [Derived] Nordeng J, Schandiz H, Solheim S, Akra S, Hoffman P, Roald B, Bendz B, Arnesen H, Helseth R, Seljeflot I. TIMP-1 expression in coronary thrombi associate with myocardial injury in ST-elevation myocardial infarction patients. Coron Artery Dis. 2022 Sep 1;33(6):446-455. doi: 10.1097/MCA.0000000000001128. Epub 2022 Jan 31. PMID 35102064
- [Derived] Nordeng J, Schandiz H, Solheim S, Akra S, Hoffman P, Roald B, Bendz B, Arnesen H, Helseth R, Seljeflot I. The Inflammasome Signaling Pathway Is Actively Regulated and Related to Myocardial Damage in Coronary Thrombi from Patients with STEMI. Mediators Inflamm. 2021 May 27;2021:5525917. doi: 10.1155/2021/5525917. eCollection 2021. PMID 34135690